CLINICAL TRIAL: NCT06989814
Title: Smart Measurement of Circulating Tumor DNA: a Tumor-agnostic Computational Tool to Improve Colorectal Cancer Care
Brief Title: Smart Measurement of Circulating Tumor DNA
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Lotte van Leeuwen, PhD Candidate, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NL87476.078.24; 14976 (Other Grant/Funding Number: KWF Kankerbestrijding)
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Neoplasms; Colorectal Neoplasms Malignant; Colorectal Neoplasms, Hereditary Nonpolyposis; Hereditary Nonpolyposis Colon Cancer
Keywords: Liquid Biopsy; Colorectal cancer; Early detection; Prevention; Surveillance; Screening
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Hematologic Tests; Blood Specimen Collection; Liquid Biopsy

STUDY DESIGN:
Intervention Model Description: Case-control study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lynch-carriers with a (colorectal) tumor (Experimental): People with a newly diagnosed Lynch-associated tumor will be asked to undergo an extra blood test.
  Interventions: Diagnostic Test: Blood Product

INTERVENTIONS:
Diagnostic Test: Blood Product — An (extra) blood test will be done on participants. This will be analyzed for circulating tumor DNA (ctDNA) via a multi-omics approach.
  Other Names: Blood test; Blood draw; Liquid biopsy

SUMMARY:
The goal of this study is to develop a blood-test which can detect colorectal cancer in early stages.

Participants will be asked to take an extra blood test, which will be analyzed further in the lab.

DETAILED DESCRIPTION:
Lynch Syndrome (LS) carriers have a predisposition to develop various types of cancer, especially colorectal cancer (CRC) and endometrial cancer (EC). LS patients are advised to undergo surveillance by colonoscopy every 2 year and gynaecological surveillance. This surveillance is deemed burdensome and fails to detect a small part of the developing CRCs and the majority of extra-colonic cancers. To ensure prevention and early detection of cancer, a reliable and accessible test is needed. Recent studies have shown the potential of the detection of tumor-derived DNA fragments (circulating tumor DNA; ctDNA). Various molecular characteristics can be used to discriminate ctDNA from healthy circulating cell-free DNA. Current ctDNA assays with the highest sensitivity and specificity to detect for example minimal residual disease (MRD) after surgery are mostly tumor-informed, which means prior information is needed from the tumor tissue about the molecular alterations present.

As this information is not available for the detection of newly arising tumors, the aim of this study is to evaluate the use of an optimized combination of tumor agnostic ctDNA characteristics for the detection of newly developing tumors.

ELIGIBILITY:
Inclusion Criteria:

(suspect) Lynch Syndrome carriers who:

* Have proven Lynch Syndrome (MMR-gene or EPCAM mutation), or have a proven microsatellite instability high (MSI-H)tumor;
* Are at least 18 years old; Have been diagnosed with any form of cancer at the time of inclusion, but have had no treatment yet;
* Have granted informed consent to participate in this study.

Exclusion Criteria:

(suspect) Lynch Syndrome carriers who:

* Are unwilling to undergo extra blood sampling;
* Are under the age of 18;
* Have no newly diagnosed tumors at time of inclusion;
* Have been treated for their tumor at time of inclusion;
* Are not able to read or understand Dutch language or are mentally not capable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Estimated ctDNA fractions in blood | Measurement at baseline
  ctDNA presence will be measured against a (presently not specified) threshold, creating a divide between 'detectable' and 'non-detectable'.
Tumor pathology | Measurement at baseline
  Tumor pathology will be revised to later compare with estimated ctDNA presence.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Wagner, Dr., Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No
Participant data will be pseudonymized for privacy purposes. Also, data will be interpreted in group form, individual patients will not receive any results on individual level.

REFERENCES:
- [Background] Mouliere F, Chandrananda D, Piskorz AM, Moore EK, Morris J, Ahlborn LB, Mair R, Goranova T, Marass F, Heider K, Wan JCM, Supernat A, Hudecova I, Gounaris I, Ros S, Jimenez-Linan M, Garcia-Corbacho J, Patel K, Ostrup O, Murphy S, Eldridge MD, Gale D, Stewart GD, Burge J, Cooper WN, van der Heijden MS, Massie CE, Watts C, Corrie P, Pacey S, Brindle KM, Baird RD, Mau-Sorensen M, Parkinson CA, Smith CG, Brenton JD, Rosenfeld N. Enhanced detection of circulating tumor DNA by fragment size analysis. Sci Transl Med. 2018 Nov 7;10(466):eaat4921. doi: 10.1126/scitranslmed.aat4921. PMID 30404863
- [Background] Deger T, Boers RG, de Weerd V, Angus L, van der Put MMJ, Boers JB, Azmani Z, van IJcken WFJ, Grunhagen DJ, van Dessel LF, Lolkema MPJK, Verhoef C, Sleijfer S, Martens JWM, Gribnau J, Wilting SM. High-throughput and affordable genome-wide methylation profiling of circulating cell-free DNA by methylated DNA sequencing (MeD-seq) of LpnPI digested fragments. Clin Epigenetics. 2021 Oct 20;13(1):196. doi: 10.1186/s13148-021-01177-4. PMID 34670587
- [Background] Schrag D, Beer TM, McDonnell CH 3rd, Nadauld L, Dilaveri CA, Reid R, Marinac CR, Chung KC, Lopatin M, Fung ET, Klein EA. Blood-based tests for multicancer early detection (PATHFINDER): a prospective cohort study. Lancet. 2023 Oct 7;402(10409):1251-1260. doi: 10.1016/S0140-6736(23)01700-2. PMID 37805216
- [Result] Eikenboom EL, Wilting SM, Deger T, Srebniak MI, Van Veghel-Plandsoen M, Boers RG, Boers JB, van IJcken WFJ, Gribnau JH, Atmodimedjo P, Dubbink HJ, Martens JWM, Spaander MCW, Wagner A. Liquid Biopsies for Colorectal Cancer and Advanced Adenoma Screening and Surveillance: What to Measure? Cancers (Basel). 2023 Sep 17;15(18):4607. doi: 10.3390/cancers15184607. PMID 37760576
- See also: Information (in Dutch) on the Dutch Cancer Society website — https://www.kwf.nl/onderzoek/onderzoeksdatabase/het-vinden-van-de-slimste-bloedmeting-voor-vroege-detectie-van-nieuwe

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT06989814/Prot_SAP_000.pdf